CLINICAL TRIAL: NCT03946969
Title: Safety and Efficacy of Combination of Sintilimab and Platinum-based Chemotherapy in Neoadjuvant Treatment of Potentially Resectable Esophageal Cancer: An Open-lable, Single-arm, Exploratory Clinical Study
Brief Title: Sintilimab in Combination With Chemotherapy in Neoadjuvant Treatment of Potentially Resectable Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Gu Yanhong, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 03
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant; Esophageal Cancer; PD-1
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — sintilimab; Cisplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab + Liposomal Paclitaxel + Cisplatin + S-1 (Experimental): Sintilimab will be administered prior to the chemotherapy in an interval of half an hour.
  Interventions: Drug: Sintilimab; Drug: Liposomal Paclitaxel + Cisplatin + S-1

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (200mg) will be given intravenously on day 1 in 3-week cycles for two cycles.
  Other Names: IBI308
Drug: Liposomal Paclitaxel + Cisplatin + S-1 — Liposomal Paclitaxel (135mg/m2), ivd, d1 + Cisplatin (25mg/m2), ivd, d1-3 + S-1 capsule (40mg), po, d1-14, repeated every 3 weeks for two cycles.
  Other Names: PFC

SUMMARY:
This study aims to investigate the safety and efficacy of sintilimab combined with platinum-based chemotherapy in neoadjuvant treatment of potentially resectable esophageal cancer.

DETAILED DESCRIPTION:
This study was designed as an open-lable, single-arm, exploratory clinical study. Sintilimab in combination with liposomal paclitaxel, cisplatin and S-1 will be given every 3 weeks to our patients for 2 cycles as neoadjuvant therapy. A radical dissection is scheduled within 6 weeks after last neoadjuvant treatment. This study will be devided for 3 phases: safety run-in, efficacy pilot and efficacy confirmation.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed esophageal squamous cell carcinoma.

The tumor is located in the middle or lower third of the esophagus ( more than 18cm below incisor), potentially resectable and requiring neoadjuvant therapy (T1b-3, Nany, M0 or T4a, N0-1, M0).

No prior treatment for this disease.

Eastern cooperative oncology group (ECOG) performance status of 0 to 1.

Adequate bone marrow, liver, cardiac and renal function as assessed by the laboratory required by protocol.

Understand and voluntarily sign the informed consent(s).

Patients who are able to complete the treatment and follow-up according to the study plan.

Patients who have sufficient tissue samples and agree to provide their tissue samples and blood samples for detailed analysis.

Female patients in child bearing period must have evidence of negative pregnancy test and agree to take effective contraceptive measures during the study.

Exclusion Criteria:

Patients who may develop tracheoesophageal fistula or aortoesophageal fistula.

Patients suffering from severe malnutrition or needing tube feeding.

Uncured patients with other malignancies within 2 years.

Patients who have active autoimmune diseases or patients who are undergoing treatment of autoimmune diseases.

Patients who need systemic glucocorticosteroid treatment (more than 10mg prednisone daily or other equivalent drugs) within 7 days before the neoadjuvant therapy or other immunosuppressive drugs.

Patients who have immune deficiency.

Patients with active viral or bacterial infection who need systemic treatment within 7 days before the neoadjuvant therapy.

Patients with uncontrolled diabetes mellitus.

Patients with interstitial pulmonary disease, noninfectious pneumonia, or pulmonary fibrosis.

Patients with preexisting symptoms of sensory or motor nerve damage (greater than Grade 1, WHO) .

Patients who have received allogeneic organ or stem cell transplants.

Patients who are allergic to drugs or related ingredients in this study.

Patients who take part in clinical trials of other drugs or biological therapy at present.

Patients with any serious or unstable medical condition or mental illness.

Patients who are dependent on or addicted to alcohol or drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility | 20 months
  Safety is defined as the incidence of Grade 3-4 Treatment-Related Adverse Events (TRAEs) from the day of neoadjuvant therapy to 30 days after surgery or within 90 days after last neoadjuvant treatment. Feasibility of surgery is defined as the incidence of TRAEs causing surgery delay of ≥30 days and/or inoperable patients.

SECONDARY OUTCOMES:
MPR rate | 20 months
  Major Pathological Response (MPR) is defined as the presence of 10% or fewer viable cancer cells in the hematoxylin and eosin (H&E)-stained slides from the resected tumor following neoadjuvant treatment.
R0 resection rate | 20 months
  R0 resection is defined as no cancer cells are seen microscopically at the resection margin following surgery.
Recurrence-Free Survival (RFS) | 5 years
  Recurrence-Free Survival (RFS) is calculated from surgery to the date of recurrence or death.
Overall Survival (OS) | 5 years
  Overall Survival (OS) is calculated from the beginning of neoadjuvant treatment to the date of death from any cause.

OTHER OUTCOMES:
Exploratory Outcomes | 20 months
  Correlation between biomarkers, including tumor mutational burden (TMB), clonal mutations, genetic alterations, and circulating tumor DNA (ctDNA), and therapeutic response to neoadjuvant therapy will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Gu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Xu X, Wang D, Liu J, Sun J, Lu M, Wang R, Hui B, Li X, Zhou C, Wang M, Qiu T, Cui S, Sun N, Li Y, Wang F, Liu C, Shao Y, Luo J, Gu Y. Neoadjuvant sintilimab and chemotherapy in patients with potentially resectable esophageal squamous cell carcinoma (KEEP-G 03): an open-label, single-arm, phase 2 trial. J Immunother Cancer. 2023 Feb;11(2):e005830. doi: 10.1136/jitc-2022-005830. PMID 36759013